CLINICAL TRIAL: NCT03944590
Title: Radiological and Clinical Outcome After Screw Osteosynthesis of Radial Head Fractures
Acronym: RadioHead
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00282; ch19Rikli
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Radial Head Fractures
Keywords: screw osteosynthesis; rupture of the interosseous membrane; collateral ligaments
MeSH Terms: conditions — Radial Head and Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient survey — patient survey on clinical outcome after screw osteosynthesis of radial head fractures
Other: analysis of radiographs — analysis of radiographs on radiological outcome after screw osteosynthesis of radial head fractures

SUMMARY:
This cohort study investigates radiological and clinical outcome after screw osteosynthesis of radial head fractures with associated injuries (such as rupture of the interosseous membrane and collateral ligaments). Interpretation of radiographs 3 and 9 months post- surgery and patient surveys will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* screw osteosynthesis of radial head fractures

Exclusion Criteria:

* unable to give consent
* dementia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing screw osteosynthesis of radial head fractures at Universitätsspital Basel between June 2010 until June 2016
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change in status of bone healing assessed by radiographs | 3 months and 9 months post surgery
  Analysis of radiographs with regard to bone healing (cortical bone, dislocation of fracture and dislocation of screws)

SECONDARY OUTCOMES:
elbow status assessed by Mayo Elbow Score (MEPS) | single time point, assessment 2 to 7 years after surgery
  A clinician-completed scoring system used to evaluate the level of disability in the elbow, assessing pain, functional status (based on number tasks performed), range of motion and joint stability. Clinical information is rated based on a 100 points scale:
  <60 - poor 60-74 - fair 75-89 - good 90-100 - excellent
Patient reported outcome of elbow surgery assessed by Oxford Elbow Score (OES) | single time point, assessment 2 to 7 years after surgery
  The Oxford Elbow Score has 12 items (questions) with 5 response options each. Each item response is scored 0 to 4, with 0 representing greater severity. Underlying the 12 items are 3 domains (sub-scales): Elbow pain, Elbow function and Social-psychological domain. Scores for each domain are calculated as the sum of each individual item score within that domain, which is then converted to a metric of 0 - 100 (lower score representing greater severity).
Patient reported outcome assessed by Quick Dash | single time point, assessment 2 to 7 years after surgery
  Quick Dash is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity level/ function level. Scoring ranges from 1 = no difficulty to 5 = unable to do. A higher score indicates a greater level of disability and severity.
Assessment on employment | single time point, assessment 2 to 7 years after surgery
  Assessment whether the patient is able to perform the original job activity as before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rikli, Prof. Dr., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland